CLINICAL TRIAL: NCT01305954
Title: LCCC 1027: Expression Of P16INK4a As A Predictor Of Myelosuppression In Patients With Breast Cancer
Brief Title: Study of the P16 Gene as a Predictor of Myelosuppression in Breast Cancer Patients
Status: Completed | Type: Observational
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: LCCC1027; 10-2121 (Other: UNC Office of Human Research Ethics)
Record Dates: First submitted 2011-02-17; First posted 2011-03-01 (Estimated); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Breast Cancer
Keywords: Breast; Cancer; Breast Cancer; New Diagnosis; Treatment; Chemotherapy; Blood; Blood Draw; Lab Draw; Gene; Gene Therapy; Geriatric; Oncology; Muss; UNC; North Carolina Cancer Hospital; Initial Treatment; CBC
MeSH Terms: conditions — Breast Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The primary purpose of this study is to measure the association between baseline expression of the senescence effector protein p16INK4a and myelosuppression due to chemotherapy in patients with breast cancer. Patients with Stage I-IV breast cancer will be included and myelosuppression will be assessed after the first cycle of chemotherapy via measurement of an absolute neutrophil count (ANC) measured one time between days 7-11 post cycle one. Study subjects will also be asked to complete a brief health behaviors questionnaire to gather information on other relevant variables.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age;
* Histologically confirmed Stage I-IV breast cancer;
* ECOG Performance Status 0-3;
* Scheduled to start a new course of chemotherapy in the neo-adjuvant, adjuvant or metastatic setting for newly diagnosed or recurrent disease;
* Growth factors, e.g., filgrastim, pegfilgrastim, are allowed, but their dose and duration will be tracked.
* Absolute Lymphocyte Count (ALC) > 500 cells/μL as determined by routine CBC with differential;
* Signed, IRB approved written informed consent.

Exclusion Criteria:

* Presence of acute, active infection;
* History of clonal bone marrow disorder (i.e., myelodysplastic or myeloproliferative disorder, acute or chronic leukemia);
* Other co-morbid illness which would impair ability to participate in the study;
* Concurrent experimental therapy (Note: concurrent biologic therapy IS permitted, provided it is not experimental).
* Prior or current receipt of histone deacetylase (HDAC) inhibitors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Breast cancer patients at UNC North Carolina Cancer Hospital and other participating sights.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2010-12; Primary Completion 2014-04-03 (Actual); Study Completion 2023-09-25 (Actual)

PRIMARY OUTCOMES:
Determine if p16INK4a Expression at Baseline is Related to Nadir Neutrophil Counts in Women with Breast Cancer Receiving Chemotherapy | 24 months
  To measure and correlate baseline p16INK4a expression in subjects with stage I-IV breast cancer starting a new course of chemotherapy with a post cycle 1 chemotherapy absolute neutrophil count (ANC).

SECONDARY OUTCOMES:
Define the Association Between p16INK4a Expression and Physical Activity, Smoking and Alcohol Consumption in Women with Breast Cancer Receiving Chemotherapy | 24 months
  To explore the associations between p16INK4a expression at baseline and amount of vigorous physical activity, smoking habits, and weekly alcohol consumption.
Explore the Associations between p16INK4a Expression at Baseline and Other Chemotherapy-Related Toxicities including Nausea and Vomiting, Neuropathy, Fatigue and Other Grade 3 and 4 Toxicities | 24 Months
  To explore the associations between p16INK4a expression at baseline and other chemotherapy-related toxicities, including the maximum toxicity experienced during that course of chemotherapy.
Explore Associations between p16INK4a Expression at Baseline, Chemotherapy Regimen, and its Effect on Patient Function | 24 months
  To explore the associations between p16INK4a expression at baseline and type of chemotherapy received, co-morbidities, concomitant medications, and tumor characteristics.

CONTACTS AND LOCATIONS:
Overall Officials: Hyman Muss, MD, Principal Investigator — University of North Carolina
Locations (1):
- University of North Carolina, Chapel Hill, North Carolina, United States

REFERENCES:
- See also: The Geriatric Oncology Research Program at UNC — http://www.unclineberger.org/geriatric